CLINICAL TRIAL: NCT03261102
Title: Therapeutic Drug Monitoring Guided Early Optimization of Adalimumab in Crohn's Disease; A Randomized Open Label Study
Brief Title: TDM Guided Early Optimization of ADAL in Crohn's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: waqqas.afif (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, waqqas.afif, Dr. Waqqas Afif MD, FRCPC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-37-2017-2793
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; Drug Monitoring; Inflammatory Bowel Diseases
Keywords: IBD; Crohn; adalimumab; ADAL
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Some of the participants, care providers and investigators will eventually, in the course of the study, have knowledge of the arm they were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard clinical care (Active Comparator): Adalimumab induction as per standard clinical care:
  * Week 0: 160 mg SC
  * Week 2: 80 mg SC
  * Followed by 40 mg SC every 2 weeks' maintenance therapy
  Interventions: Biological: Adalimumab
- Active optimization (Active Comparator): Same as Standard clinical care Arm, except:
  * If ADAL trough ≤15 μg/ml, dose escalation with 80 mg SC at week 6 followed by 40 mg SC every week
  * If ADAL trough >15 μg/ml, no dose escalation and continued standard of care dosing
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab
  Other Names: Humira

SUMMARY:
To investigate the influence of early therapeutic drug monitoring and dose optimization on disease outcome in Crohn's patients treated with Adalimumab.

DETAILED DESCRIPTION:
This is an investigator initiated randomized open label study. This study is designed to compare whether increasing the dose of adalimumab based on the level the drug in the blood to a target level early in the treatment course would lead to better outcomes for patients as compared to the standard doses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Crohn's disease diagnosed based on standard objective methodology (clinical, biochemical, endoscopic, histological and radiological correlation).
* Active disease based on Harvey Bradshaw Index (HBI >5) and elevated C-reactive protein (CRP) (>normal reference range for local laboratory) OR fecal calprotectin (FCP) (>250 µg/g)
* Due to commence treatment with ADAL.

Exclusion Criteria:

* Severe co-existing cardiopulmonary, hepatic, renal, neurologic, or rheumatologic disease.
* History of active HIV, hepatitis B or C infection,
* Patients with ileostomy/colostomy, ileal-pouch anal anastomosis or severe perianal fistulising disease.
* Pregnancy
* Prior exposure to ADAL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved remission | Week 12
  Clinical remission will be scored by a Harvey-Bradshaw Index < 5 AND Biochemical remission will be scored by C-reactive protein < 5 mg/l OR Fecal calprotectin <250 μg/g (combination endpoint)

SECONDARY OUTCOMES:
Proportion of subjects who achieved clinical response | From Week 0 to Week 12
  Clinical response will be evaluated by a decreased in Harvey-Bradshaw Index score AND a decreased level of C-reactive protein OR Fecal calprotectin
Therapeutic drug monitoring | At Week 8, 12
  Adalimumab drug concentration at week 8 and 12 AND proportion of subjects with antibody to Adalimumab at Week 8 and 12 on the rate i. Clinical response/remission (HBI<5) ii. Biochemical response/remission (CRP within normal reference range) iii. Endoscopic response (SES-CD reduction of ≥50% from baseline) / remission (SES-CD ≤3)
Proportion of steroid free subjects | At Week 12
  Steroid free defined as patients being steroid free at Week 12
Subjects well-being | From Week 0 to Week 12
  Subjects well-being will be scored using the validated questionnaire Short inflammatory bowel disease questionnaire (SIBDQ)
Rates of complications | 12 weeks
  Rates of complications, including hospitalization, surgery, adverse reaction, and corticosteroid use.

CONTACTS AND LOCATIONS:
Overall Officials: Waqqas Afif, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (6):
- Canada (6):
  - University of Calgary Medical Center (UCMC), Calgary, Alberta
  - The University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre (LHSC) University Hospital, London, Ontario
  - The Ottawa Hospital, IBD Centre of Excellence, Ottawa, Ontario
  - McGill University Hospital Center (MUHC), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No